CLINICAL TRIAL: NCT00892658
Title: A Phase I Study of Sorafenib and Radiation Therapy in Patients With Hepatocellular Carcinoma
Brief Title: Sorafenib-RT in Treating Hepatocellular Carcinoma (SHEP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0761-C
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Sorafenib; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib + RT (Experimental)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Patients will receive sorafenib alone (following the dose escalation scheme) for one week, followed by 2 weeks of concurrent administration of sorafenib with conformal radiation therapy (6 fractions over two weeks). Sorafenib administration will continue for four weeks following completion of radiation. At three months following radiation, when liver toxicity is assessed, full dose sorafenib (400mg PO BID) will then be initiated and continued until disease progression or serious toxicity occurs, to a maximum time of 12 months.

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common cancers worldwide. The incidence is highest in Asia and it is increasing in North America, with a two to three fold increase in mortality in North America expected over the next two decades. Previous research has shown that tumours often have abnormal blood vessels that may reduce the effect of radiation therapy. New drugs, known as "anti-angiogenic" drugs have been shown in animal and human studies to damage or change tumour blood vessels in ways that may make tumors more sensitive to radiation treatment. 38-44 patients diagnosed with HCC will be invited to take part in this study. Upon completion, this study will establish the safety of the combination of radiation and sorafenib in patients with HCC. This will also establish preliminary data regarding efficacy of the combination and investigate potential imaging and serum/tissue markers surrogates for tumor response and/or drug activity.

DETAILED DESCRIPTION:
The study design will include 2 radiation strata of patients, with a constant radiation dose for strata 1 requiring a low volume of liver to be irradiated, and a variable dose defined based on the effective liver volume irradiated in the second strata, which will require more liver volume to be irradiated, based on our prior experience. Both stratas one and two will be accrued concurrently. Biologic response will be assessed using standard contrast CT scans. Correlative studies of biological markers, perfusion CT, and microbubble contrast enhanced ultrasound will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have HCC either

  * confirmed pathologically
  * diagnosed by showing vascular enhancement of the lesion on at least two imaging techniques
  * diagnosed by showing vascular enhancement on a single technique if the AFP is over 200, in the setting of cirrhosis or chronic hepatitis B without cirrhosis. Biopsies are mandatory (unless an absolute contraindication exists).
* The tumour must be unresectable or medically inoperable
* At least 800 cc of non-tumor liver
* Patients must be > 4 weeks since any major surgery.
* Patients may have had previous systemic treatment (with at least a 2 week break from systemic therapy to start of radiation therapy. Prior sorafenib or any other targeted therapy with anti-VEGF activity is not permitted.
* Child-Pugh Liver score A
* Barcelona-Clinic Liver Cancer (BCLC) score A or B or C (BCLC C permitted if ECOG 0-1 and Child Pugh A, with portal invasion)
* Age 18 years or older.
* Life expectancy of equal to or greater than 3 months.
* ECOG performance status 0-1.
* Patients must have normal organ and marrow function.
* Ability to understand and the willingness to sign a written informed consent document.
* Negative pregnancy test for women of child bearing age
* If the patient has a history of varices and portal hypertension, elective treatment (e.g. banding) of varices will be performed prior to start of radiation therapy.
* The effects of Sorafenib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Serious medical conditions that might be aggravated by treatment, including but not limited to: myocardial infarction within 6 months, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, active hepatitis or cerebrovascular disease with previous stroke within the past 12 months.
* Patients may not be receiving any other investigational agents concurrently or within 2 weeks of initiation of treatment.
* Pregnant women
* Patients with immune deficiency
* Ascites (on imaging or clinical exam).
* Prior liver or upper abdomen radiation therapy.
* Resectable hepatocellular carcinoma.
* Thrombolytic therapy within 4 weeks, or any concurrent anti-coagulant therapy.
* Uncontrolled hypertension
* Patients with other active malignancies
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib.
* Patients with active hepatitis or encephalopathy related to liver failure.
* Patients with any bleeding or clotting disorder.
* Patients with unhealed wounds or ulcers.
* Prior sorafenib treatment is not permitted.
* Patient with nausea and vomiting refractory to medical therapies, significant prior bowel resection, and inflammatory bowel disease.
* Patients with evidence of extrahepatic metastases
* Patients on Rifampin, St.John's Wort, Phenytonin, Carbamazepine, Phenobarbital, or chronic use (more than 4 weeks) of dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Determine the MTD of sorafenib and RT in patients with hepatocellular carcinoma using an iso-toxicity radiation dose allocation scheme. Determine the acute toxicity (< 3 months) of sorafenib when combined with RT. | 1 year enrollment; 5 years follow-up

SECONDARY OUTCOMES:
Determine late toxicities, in-field local control at 3 months, overall survival, progression time, and progression free survival. Quantify alteration in perfusion parameters.Assess serum and tissue biomarkers. Assess quality of life in these patients. | 1 year enrollment; 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital; Anthony Brade, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada